CLINICAL TRIAL: NCT02609269
Title: Prospective Expression Analysis Using The Decipher Genomics Resource for Intelligent Discovery (GRID)® and Data Sharing Program
Brief Title: Decipher Genomics Resource for Intelligent Discovery
Acronym: GRID®
Status: Enrolling by invitation | Type: Observational
Sponsor: GenomeDx Biosciences Corp (Industry)
Collaborators: Veracyte, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GRD001
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer; Bladder Cancer; Renal Cancer
Keywords: Decipher; Transcriptome; Gene Expression
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — RNA extracted from tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Decipher GRID Patients: Patients who have been tested with any of the Decipher clinical tests
  Interventions: Other: Decipher Cancer Classifier

INTERVENTIONS:
Other: Decipher Cancer Classifier — The Decipher are gene expression-based tests that are used to better risk stratify or characterize tumor biology that are commercially available through Veracyte, Inc CLIA & CAP certified laboratory in San Diego, CA
  Other Names: Decipher Biopsy, Decipher RP, Decipher Bladder, Decipher Renal, Decipher Test

SUMMARY:
To prospectively evaluate the utility of genomic expression data as a tool to better characterize the tumors of individual patients, and to understand how genomic information from individual patients undergoing routine clinical testing can be used in population-level analysis to improve treatment and outcomes.

DETAILED DESCRIPTION:
Observational study involving the release of tumor genome-wide expression data generated by the Decipher assay which will be linked to clinical treatment and outcome data for patients in whom Decipher clinical testing was performed. The GRID database population will be used to characterize the genomics of cancer and discover or validate gene expression signatures that may be useful for understanding of the biology of the disease and implementing precision medicine approaches for cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects that have had a Decipher clinical test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing Decipher testing in the clinical setting. It is understood that the Decipher test results may be used as a part of normal clinical care. Any patient meeting the following criteria who has been tested with Decipher can participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Link complete genomic RNA expression array data generated from Decipher testing with clinical data for patients who consent to participate. | Through study completion, an average of 1 year
  Role of genomic expression data in the biology of certain cancers

CONTACTS AND LOCATIONS:
Overall Officials: Elai Davicioni, PhD, Principal Investigator — Veracyte, Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karnes RJ, Bergstralh EJ, Davicioni E, Ghadessi M, Buerki C, Mitra AP, Crisan A, Erho N, Vergara IA, Lam LL, Carlson R, Thompson DJ, Haddad Z, Zimmermann B, Sierocinski T, Triche TJ, Kollmeyer T, Ballman KV, Black PC, Klee GG, Jenkins RB. Validation of a genomic classifier that predicts metastasis following radical prostatectomy in an at risk patient population. J Urol. 2013 Dec;190(6):2047-53. doi: 10.1016/j.juro.2013.06.017. Epub 2013 Jun 11. PMID 23770138
- [Background] Ross AE, Johnson MH, Yousefi K, Davicioni E, Netto GJ, Marchionni L, Fedor HL, Glavaris S, Choeurng V, Buerki C, Erho N, Lam LL, Humphreys EB, Faraj S, Bezerra SM, Han M, Partin AW, Trock BJ, Schaeffer EM. Tissue-based Genomics Augments Post-prostatectomy Risk Stratification in a Natural History Cohort of Intermediate- and High-Risk Men. Eur Urol. 2016 Jan;69(1):157-65. doi: 10.1016/j.eururo.2015.05.042. Epub 2015 Jun 6. PMID 26058959
- [Background] Cooperberg MR, Davicioni E, Crisan A, Jenkins RB, Ghadessi M, Karnes RJ. Combined value of validated clinical and genomic risk stratification tools for predicting prostate cancer mortality in a high-risk prostatectomy cohort. Eur Urol. 2015 Feb;67(2):326-33. doi: 10.1016/j.eururo.2014.05.039. Epub 2014 Jul 2. PMID 24998118
- [Background] Den RB, Yousefi K, Trabulsi EJ, Abdollah F, Choeurng V, Feng FY, Dicker AP, Lallas CD, Gomella LG, Davicioni E, Karnes RJ. Genomic classifier identifies men with adverse pathology after radical prostatectomy who benefit from adjuvant radiation therapy. J Clin Oncol. 2015 Mar 10;33(8):944-51. doi: 10.1200/JCO.2014.59.0026. Epub 2015 Feb 9. PMID 25667284
- [Background] Den RB, Feng FY, Showalter TN, Mishra MV, Trabulsi EJ, Lallas CD, Gomella LG, Kelly WK, Birbe RC, McCue PA, Ghadessi M, Yousefi K, Davicioni E, Knudsen KE, Dicker AP. Genomic prostate cancer classifier predicts biochemical failure and metastases in patients after postoperative radiation therapy. Int J Radiat Oncol Biol Phys. 2014 Aug 1;89(5):1038-1046. doi: 10.1016/j.ijrobp.2014.04.052. Epub 2014 Jul 8. PMID 25035207
- [Background] Erho N, Crisan A, Vergara IA, Mitra AP, Ghadessi M, Buerki C, Bergstralh EJ, Kollmeyer T, Fink S, Haddad Z, Zimmermann B, Sierocinski T, Ballman KV, Triche TJ, Black PC, Karnes RJ, Klee G, Davicioni E, Jenkins RB. Discovery and validation of a prostate cancer genomic classifier that predicts early metastasis following radical prostatectomy. PLoS One. 2013 Jun 24;8(6):e66855. doi: 10.1371/journal.pone.0066855. Print 2013. PMID 23826159
- [Background] Jairath NK, Dal Pra A, Vince R Jr, Dess RT, Jackson WC, Tosoian JJ, McBride SM, Zhao SG, Berlin A, Mahal BA, Kishan AU, Den RB, Freedland SJ, Salami SS, Kaffenberger SD, Pollack A, Tran P, Mehra R, Morgan TM, Weiner AB, Mohamad O, Carroll PR, Cooperberg MR, Karnes RJ, Nguyen PL, Michalski JM, Tward JD, Feng FY, Schaeffer EM, Spratt DE. A Systematic Review of the Evidence for the Decipher Genomic Classifier in Prostate Cancer. Eur Urol. 2021 Mar;79(3):374-383. doi: 10.1016/j.eururo.2020.11.021. Epub 2020 Dec 5. PMID 33293078
- [Background] Qiu X, Boufaied N, Hallal T, Feit A, de Polo A, Luoma AM, Alahmadi W, Larocque J, Zadra G, Xie Y, Gu S, Tang Q, Zhang Y, Syamala S, Seo JH, Bell C, O'Connor E, Liu Y, Schaeffer EM, Jeffrey Karnes R, Weinmann S, Davicioni E, Morrissey C, Cejas P, Ellis L, Loda M, Wucherpfennig KW, Pomerantz MM, Spratt DE, Corey E, Freedman ML, Shirley Liu X, Brown M, Long HW, Labbe DP. MYC drives aggressive prostate cancer by disrupting transcriptional pause release at androgen receptor targets. Nat Commun. 2022 May 13;13(1):2559. doi: 10.1038/s41467-022-30257-z. PMID 35562350
- [Background] Zhao SG, Chang SL, Erho N, Yu M, Lehrer J, Alshalalfa M, Speers C, Cooperberg MR, Kim W, Ryan CJ, Den RB, Freedland SJ, Posadas E, Sandler H, Klein EA, Black P, Seiler R, Tomlins SA, Chinnaiyan AM, Jenkins RB, Davicioni E, Ross AE, Schaeffer EM, Nguyen PL, Carroll PR, Karnes RJ, Spratt DE, Feng FY. Associations of Luminal and Basal Subtyping of Prostate Cancer With Prognosis and Response to Androgen Deprivation Therapy. JAMA Oncol. 2017 Dec 1;3(12):1663-1672. doi: 10.1001/jamaoncol.2017.0751. PMID 28494073
- [Background] Feng FY, Huang HC, Spratt DE, Zhao SG, Sandler HM, Simko JP, Davicioni E, Nguyen PL, Pollack A, Efstathiou JA, Dicker AP, Todorovic T, Margrave J, Liu YS, Dabbas B, Thompson DJS, Das R, Dignam JJ, Sweeney C, Attard G, Bahary JP, Lukka HR, Hall WA, Pisansky TM, Shah AB, Pugh SL, Shipley WU, Tran PT. Validation of a 22-Gene Genomic Classifier in Patients With Recurrent Prostate Cancer: An Ancillary Study of the NRG/RTOG 9601 Randomized Clinical Trial. JAMA Oncol. 2021 Apr 1;7(4):544-552. doi: 10.1001/jamaoncol.2020.7671. PMID 33570548
- [Result] Adams EJ, Karthaus WR, Hoover E, Liu D, Gruet A, Zhang Z, Cho H, DiLoreto R, Chhangawala S, Liu Y, Watson PA, Davicioni E, Sboner A, Barbieri CE, Bose R, Leslie CS, Sawyers CL. FOXA1 mutations alter pioneering activity, differentiation and prostate cancer phenotypes. Nature. 2019 Jul;571(7765):408-412. doi: 10.1038/s41586-019-1318-9. Epub 2019 Jun 26. PMID 31243370
- [Result] Mahal BA, Yang DD, Wang NQ, Alshalalfa M, Davicioni E, Choeurng V, Schaeffer EM, Ross AE, Spratt DE, Den RB, Martin NE, Mouw KW, Orio PF 3rd, Choueiri TK, Taplin ME, Trinh QD, Feng FY, Nguyen PL. Clinical and Genomic Characterization of Low-Prostate-specific Antigen, High-grade Prostate Cancer. Eur Urol. 2018 Aug;74(2):146-154. doi: 10.1016/j.eururo.2018.01.043. Epub 2018 Feb 22. PMID 29478736
- [Result] Chu CE, Alshalalfa M, Sjostrom M, Zhao SG, Liu Y, Chou J, Herlemann A, Mahal B, Kishan AU, Spratt DE, Cooperberg M, Small E, Wong A, Porten S, Hope TA, Ross AE, Davicioni E, Nguyen P, Karnes RJ, Carroll PR, Schaeffer E, Feng FY. Prostate-specific Membrane Antigen and Fluciclovine Transporter Genes are Associated with Variable Clinical Features and Molecular Subtypes of Primary Prostate Cancer. Eur Urol. 2021 Jun;79(6):717-721. doi: 10.1016/j.eururo.2021.03.017. Epub 2021 Apr 8. PMID 33840559
- [Result] Kensler KH, Awasthi S, Alshalalfa M, Trock BJ, Freedland SJ, Freeman MR, You S, Mahal BA, Den RB, Dicker AP, Karnes RJ, Klein EA, Lal P, Liu Y, Davicioni E, Rayford W, Yamoah K, Rebbeck TR. Variation in Molecularly Defined Prostate Tumor Subtypes by Self-identified Race. Eur Urol Open Sci. 2022 Apr 26;40:19-26. doi: 10.1016/j.euros.2022.03.014. eCollection 2022 Jun. PMID 35638091
- [Result] Zhao SG, Lehrer J, Chang SL, Das R, Erho N, Liu Y, Sjostrom M, Den RB, Freedland SJ, Klein EA, Karnes RJ, Schaeffer EM, Xu M, Speers C, Nguyen PL, Ross AE, Chan JM, Cooperberg MR, Carroll PR, Davicioni E, Fong L, Spratt DE, Feng FY. The Immune Landscape of Prostate Cancer and Nomination of PD-L2 as a Potential Therapeutic Target. J Natl Cancer Inst. 2019 Mar 1;111(3):301-310. doi: 10.1093/jnci/djy141. PMID 30321406
- [Result] Cooperberg MR, Erho N, Chan JM, Feng FY, Fishbane N, Zhao SG, Simko JP, Cowan JE, Lehrer J, Alshalalfa M, Kolisnik T, Chelliserry J, Margrave J, Aranes M, Plessis MD, Buerki C, Tenggara I, Davicioni E, Carroll PR. The Diverse Genomic Landscape of Clinically Low-risk Prostate Cancer. Eur Urol. 2018 Oct;74(4):444-452. doi: 10.1016/j.eururo.2018.05.014. Epub 2018 May 28. PMID 29853306
- [Result] Rayford W, Beksac AT, Alger J, Alshalalfa M, Ahmed M, Khan I, Falagario UG, Liu Y, Davicioni E, Spratt DE, Schaeffer EM, Feng FY, Mahal B, Nguyen PL, Den RB, Greenberger MD, Bradley R, Watson JM, Beamer M, Stamatakis L, Carmen DJ, Awasthi S, Hwang J, Weil R, Merisaari H, Mohamed N, Deane LA, Chakravarty D, Yadav KK, Yamoah K, Nair SS, Tewari AK. Comparative analysis of 1152 African-American and European-American men with prostate cancer identifies distinct genomic and immunological differences. Commun Biol. 2021 Jun 3;4(1):670. doi: 10.1038/s42003-021-02140-y. PMID 34083737
- [Result] Spratt DE, Zhang J, Santiago-Jimenez M, Dess RT, Davis JW, Den RB, Dicker AP, Kane CJ, Pollack A, Stoyanova R, Abdollah F, Ross AE, Cole A, Uchio E, Randall JM, Nguyen H, Zhao SG, Mehra R, Glass AG, Lam LLC, Chelliserry J, du Plessis M, Choeurng V, Aranes M, Kolisnik T, Margrave J, Alter J, Jordan J, Buerki C, Yousefi K, Haddad Z, Davicioni E, Trabulsi EJ, Loeb S, Tewari A, Carroll PR, Weinmann S, Schaeffer EM, Klein EA, Karnes RJ, Feng FY, Nguyen PL. Development and Validation of a Novel Integrated Clinical-Genomic Risk Group Classification for Localized Prostate Cancer. J Clin Oncol. 2018 Feb 20;36(6):581-590. doi: 10.1200/JCO.2017.74.2940. Epub 2017 Nov 29. PMID 29185869
- [Result] Muralidhar V, Zhang J, Wang Q, Mahal BA, Butler SS, Spratt DE, Davicioni E, Sartor O, Feng FY, Mouw KW, Nguyen PL. Genomic Validation of 3-Tiered Clinical Subclassification of High-Risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2019 Nov 1;105(3):621-627. doi: 10.1016/j.ijrobp.2019.06.2510. Epub 2019 Jul 2. PMID 31271825
- [Result] Zhao SG, Evans JR, Kothari V, Sun G, Larm A, Mondine V, Schaeffer EM, Ross AE, Klein EA, Den RB, Dicker AP, Karnes RJ, Erho N, Nguyen PL, Davicioni E, Feng FY. The Landscape of Prognostic Outlier Genes in High-Risk Prostate Cancer. Clin Cancer Res. 2016 Apr 1;22(7):1777-86. doi: 10.1158/1078-0432.CCR-15-1250. Epub 2015 Dec 2. PMID 26631616
- [Result] Chipidza FE, Alshalalfa M, Mahal BA, Karnes RJ, Liu Y, Davicioni E, Martin NE, Mouw KW, Feng FY, Nguyen PL, Muralidhar V. Development and Validation of a Novel TP53 Mutation Signature That Predicts Risk of Metastasis in Primary Prostate Cancer. Clin Genitourin Cancer. 2021 Jun;19(3):246-254.e5. doi: 10.1016/j.clgc.2020.08.004. Epub 2020 Aug 13. PMID 32896505
- [Result] Goldberg H, Spratt D, Chandrasekar T, Klaassen Z, Wallis CJD, Santiago-Jimenez M, Fishbane N, Davicioni E, Noorani R, Ahmad AE, Herrera Caceres JO, Alibhai S, Berlin A, Fleshner NE. Clinical-genomic Characterization Unveils More Aggressive Disease Features in Elderly Prostate Cancer Patients with Low-grade Disease. Eur Urol Focus. 2021 Jul;7(4):797-806. doi: 10.1016/j.euf.2020.02.008. Epub 2020 Mar 7. PMID 32156491
- [Result] Kishan AU, Romero T, Alshalalfa M, Liu Y, Tran PT, Nickols NG, Ye H, Sajed D, Rettig MB, Reiter RE, Garraway IP, Spratt DE, Freedland SJ, Zhao X, Li Z, Deek M, Livingstone J, Mahal BA, Nguyen PL, Feng FY, Den RB, Schaeffer EM, Lotan TL, Karnes RJ, Klein EA, Ross AE, Grogan T, Davicioni E, Elashoff D, Boutros PC, Weidhaas JB. Transcriptomic Heterogeneity of Gleason Grade Group 5 Prostate Cancer. Eur Urol. 2020 Sep;78(3):327-332. doi: 10.1016/j.eururo.2020.05.009. Epub 2020 May 24. PMID 32461072
- [Derived] Hall WA, Fishbane N, Liu Y, Xu MJ, Davicioni E, Mahal BA, Den RB, Dess RT, Jackson WC, Wong AC, Schaeffer EM, Karnes RJ, Carroll PR, Cooperberg MR, Bismar TA, Kim HL, Klein EA, Davis JW, Ross AE, Tosoian JJ, Morgan TM, Mehra R, Salami SS, Nguyen PL, Lawton CAF, Spratt DE, Feng F. Development and Validation of a Genomic Tool to Predict Seminal Vesicle Invasion in Adenocarcinoma of the Prostate. JCO Precis Oncol. 2020 Nov;4:1228-1238. doi: 10.1200/PO.20.00013. PMID 35050780
- [Derived] Berglund AE, Rounbehler RJ, Gerke T, Awasthi S, Cheng CH, Takhar M, Davicioni E, Alshalalfa M, Erho N, Klein EA, Freedland SJ, Ross AE, Schaeffer EM, Trock BJ, Den RB, Cleveland JL, Park JY, Dhillon J, Yamoah K. Distinct transcriptional repertoire of the androgen receptor in ETS fusion-negative prostate cancer. Prostate Cancer Prostatic Dis. 2019 May;22(2):292-302. doi: 10.1038/s41391-018-0103-4. Epub 2018 Oct 26. PMID 30367117
- See also: Website for Decipher GRID — https://decipherbio.com/grid/
- See also: Website for Decipher by Veracyte (study sponsor) — http://www.decipherbio.com